CLINICAL TRIAL: NCT07310771
Title: A Single-Arm Phase II Study of Sintilimab Plus Nimotuzumab and Chemotherapy Followed by Definitive Chemoradiotherapy With Nimotuzumab for Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Sintilimab-Nimotuzumab Induction Followed by Chemoradiation-Nimotuzumab in LA-HNSCC: Single-Arm Phase II
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K2025-193-01
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Locally Advanced Head and Neck Squamous Cell Carcinoma (LA-SCCHN)
MeSH Terms: interventions — Drug Therapy; nimotuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab combined with chemotherapy and nimotuzumab for patients with LA-SCCHN (Experimental)
  Interventions: Drug: Sintilimab combined with chemotherapy and nimotuzumab

INTERVENTIONS:
Drug: Sintilimab combined with chemotherapy and nimotuzumab — The study plans to enroll patients with locally advanced squamous cell carcinoma of the head and neck. After induction with sintilimab plus paclitaxel, cisplatin, and nimotuzumab, participants will receive concurrent chemoradiotherapy with nimotuzumab, followed by maintenance sintilimab monotherapy until disease progression, unacceptable toxicity, death, or withdrawal of consent.

SUMMARY:
Although multiple immune-checkpoint inhibitors (ICIs) have demonstrated efficacy in recurrent or metastatic squamous-cell carcinoma of the head and neck (R/M-SCCHN), outcomes in the locally advanced (LA-SCCHN) setting remain suboptimal, and treatment continues to pose a major therapeutic challenge. Incremental improvements in efficacy are still required, necessitating the development of more effective regimens. Whether combining an ICI with chemotherapy and nimotuzumab can confer additional clinical benefit in LA-SCCHN remains to be determined. Against this backdrop, we designed a single-arm, phase II, single-centre clinical trial to evaluate the efficacy and safety of sintilimab plus chemotherapy and nimotuzumab for patients with LA-SCCHN.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent, with full understanding of and agreement to comply with study requirements and the visit schedule.
2. Age 18-75 years (inclusive) at the time of informed consent; either sex.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
4. Histologically or cytologically confirmed stage III-IVB squamous cell carcinoma of the head and neck as assessed by the investigator.
5. Documented EGFR-positive tumor.
6. No prior systemic therapy for head and neck squamous cell carcinoma.
7. At least one measurable lesion per RECIST v1.1.
8. Estimated life expectancy ≥ 12 weeks.
9. Adequate bone-marrow and organ function.

Exclusion Criteria:

1. Known hypersensitivity to any component of PD(L)-1 inhibitors, paclitaxel, or cisplatin.
2. Prior or concurrent malignancy (except adequately treated basal-cell carcinoma, cervical carcinoma in situ, or papillary thyroid carcinoma disease-free for >5 years).
3. Uncontrolled cardiac symptoms or clinically significant cardiac disease.
4. Previous therapy with anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibodies, or receipt of therapeutic cancer vaccines or live vaccines within 4 weeks before first study-dose administration.
5. Failure to recover to ≤ Grade 1 (per CTCAE) from prior anti-tumour therapy-except alopecia or residual neurotoxicity related to prior platinum-before first study dose.
6. Severe infection (> CTCAE Grade 2) within 4 weeks before first study dose.
7. Active autoimmune disease or documented autoimmune-disease history requiring systemic therapy.
8. History of immunodeficiency, including positive HIV test, congenital or acquired immunodeficiency syndromes, or prior solid-organ or allogeneic bone-marrow transplantation.
9. History of interstitial lung disease or non-infectious pneumonitis.
10. Evidence of active tuberculosis infection on history or CT imaging.
11. Active hepatitis B (HBV DNA ≥ 500 IU/mL or ≥ 2,500 copies/mL).
12. History of substance abuse, alcohol abuse, or drug addiction.
13. Pregnant or lactating women.
14. Any condition that, in the investigator's opinion, could necessitate premature withdrawal from the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2027-07-10 (Estimated); Study Completion 2029-07-10 (Estimated)

PRIMARY OUTCOMES:
Larynx-preservation rate at 3 months post-radiotherapy | 3 months

SECONDARY OUTCOMES:
objective response rate | 24 months
One-year progression-free survival (PFS) rates | 12 months
Two-year progression-free survival (PFS) rates | 24 months
One-year loco-regional relapse-free survival (LRFS) rates. | 12 months
two-year loco-regional relapse-free survival (LRFS) rates. | 24 months
One- year distant-metastasis-free survival (DMFS) rates. | 12 months
two-year distant-metastasis-free survival (DMFS) rates | 24 months
One-year larynx-preservation rates | 12 months
AE/SAE | 42 months

IPD SHARING:
Plan to Share IPD: Yes